CLINICAL TRIAL: NCT01648205
Title: Efficacy of Ranolazine in LQT3 Patients
Brief Title: Long-term Efficacy Study of Sodium Channel Blocker in LQT3 Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Wojciech Zareba, Professor of Medicine, University of Rochester
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: IN-US-259-0128
Record Dates: First submitted 2012-07-18; First posted 2012-07-24 (Estimated); Results first posted 2022-04-07 (Actual); Last update posted 2022-04-07 (Actual); Status verified 2022-03

CONDITIONS: Long QT Syndrome
Keywords: ranolazine; clinical trial
MeSH Terms: conditions — Long QT Syndrome | interventions — Ranolazine

STUDY DESIGN:
Intervention Model Description: Patients will receive placebo for 1 month and subsequently ranolazine 1000mg twice a day for 5 months.
Who Masked: Participant, Outcomes Assessor
Masking Description: Matching placebo and ranolazine pills were used. Patients were blinded regarding administration of medication. ECG Core Lab reading ECGs was blinded regarding drug assignment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Placebo followed by Ranolazine Administration (Experimental): Placebo for 1 month and Ranolazine for 5 months.
  Interventions: Drug: Placebo; Drug: Ranolazine

INTERVENTIONS:
Drug: Placebo — Matching Placebo will be given for first month.
Drug: Ranolazine — Patients will receive ranolazine 1000mg bid for subsequent 5 months.
  Other Names: Ranexa

SUMMARY:
The purpose of this study is to determine whether late sodium channel blockade might be effective in shortening the QTc interval in various LQT3 mutations and be considered as a safe therapeutic option for LQT3 patients.

DETAILED DESCRIPTION:
Long QT syndrome (LQTS) is a genetic disorder characterized by prolongation of the QT interval in the electrocardiogram (ECG) and a propensity to torsade de pointes ventricular tachycardia frequently leading to syncope, cardiac arrest, or sudden death usually in young otherwise healthy individuals. The long QT syndrome is caused by mutations of predominantly potassium and sodium ion channel genes or channel-related proteins. The most common types of LQTS affect: the slow delayed rectifier potassium repolarization channel (KCNQ1; LQT1) resulting in a reduction in IKs current; the rapid delayed rectifying potassium repolarization channel (KCNH2; LQT2) resulting in a reduction in IKr current; and the sodium channel (SCN5A; LQT3) resulting in an increase in late INa current. Among positively genotyped patients, LQT1 and LQT2 account for about 90% of LQTS cases, whereas LQT3 accounts for about 5% to 8% of cases. LQT3 patients represent a challenging cohort of patients. Unlike patients with LQT1 and LQT2 form of this disorder, the LQT3 patients have high lethality of cardiac events with 1 in 5 patients dying suddenly during their first syncopal or arrhythmic event. In childhood (age 0-18) in the analysis of 1,404 patients, LQT3 was found to be associated with significantly higher risk of aborted cardiac arrest or death than LQT1 and LQT2. A similar pattern is observed in LQTS patients after age 40 in whom LQT3 patients show the highest risk. Optimal therapy in LQT3 patients remains controversial. There are data showing that sodium current blockers including mexiletine and flecainide shorten QTc duration in LQT3 patients. Ranolazine is a selective late sodium current inhibitor that has been also showed to reduce QTc in DKPQ mutation and D1790G mutation patients. However, data on long-term effectiveness of ranolazine are limited.

This single-blinded study evaluated a long-term effects of ranolazine on QTc duration in LQT3 patients with various LQT3 mutations. Enrolled subjects are treated for 1 months with matching placebo and next for subsequent 5 months with ranolazine with ECG recorded at baseline, 1 , 2, and 6 months of follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Genotyped positive for LQT3 (SCN5A) mutation
* Age 21 years or older
* Not currently taking an antiarrhythmic drug (beta blockers are allowed)
* Enrolled in LQTS Registry

Exclusion Criteria:

* Age less than 21 years
* Not confirmed to have an LQT3 mutation
* Significant co-morbidity that would preclude subject's safe participation in this study
* Females who are pregnant or nursing
* Females of childbearing age who are not using acceptable method of birth control
* Evidence of prior sensitivity to ranolazine
* Hepatic or renal disease that might adversely affect ranolazine excretion
* Currently taking strong CYP3A inhibitors
* Currently taking P-gp inhibitors
* Currently taking CYP3A inducers
* In vitro studies of specific mutation show no effect of ranolazine on late sodium current kinetics or show repolarization prolongation

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-09; Primary Completion 2018-07-20 (Actual); Study Completion 2018-07-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wojciech Zareba, MD,PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moss AJ, Zareba W, Schwarz KQ, Rosero S, McNitt S, Robinson JL. Ranolazine shortens repolarization in patients with sustained inward sodium current due to type-3 long-QT syndrome. J Cardiovasc Electrophysiol. 2008 Dec;19(12):1289-93. doi: 10.1111/j.1540-8167.2008.01246.x. Epub 2008 Jul 25. PMID 18662191
- [Background] Zareba W, Moss AJ, Schwartz PJ, Vincent GM, Robinson JL, Priori SG, Benhorin J, Locati EH, Towbin JA, Keating MT, Lehmann MH, Hall WJ. Influence of the genotype on the clinical course of the long-QT syndrome. International Long-QT Syndrome Registry Research Group. N Engl J Med. 1998 Oct 1;339(14):960-5. doi: 10.1056/NEJM199810013391404. PMID 9753711
- [Background] Zareba W, Moss AJ, Locati EH, Lehmann MH, Peterson DR, Hall WJ, Schwartz PJ, Vincent GM, Priori SG, Benhorin J, Towbin JA, Robinson JL, Andrews ML, Napolitano C, Timothy K, Zhang L, Medina A; International Long QT Syndrome Registry. Modulating effects of age and gender on the clinical course of long QT syndrome by genotype. J Am Coll Cardiol. 2003 Jul 2;42(1):103-9. doi: 10.1016/s0735-1097(03)00554-0. PMID 12849668
- [Background] Schwartz PJ, Priori SG, Locati EH, Napolitano C, Cantu F, Towbin JA, Keating MT, Hammoude H, Brown AM, Chen LS, Colatsky TJ. Long QT syndrome patients with mutations of the SCN5A and HERG genes have differential responses to Na+ channel blockade and to increases in heart rate. Implications for gene-specific therapy. Circulation. 1995 Dec 15;92(12):3381-6. doi: 10.1161/01.cir.92.12.3381. PMID 8521555
- [Background] Benhorin J, Taub R, Goldmit M, Kerem B, Kass RS, Windman I, Medina A. Effects of flecainide in patients with new SCN5A mutation: mutation-specific therapy for long-QT syndrome? Circulation. 2000 Apr 11;101(14):1698-706. doi: 10.1161/01.cir.101.14.1698. PMID 10758053

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: There were 25 subjects enrolled receiving placebo for 1 month with ECG to be obtained at baseline and at 1 month.
Period: Placebo
Arm/Group | Placebo
Started (ECG data were available at 1 months in 21 of 25 subjects: one subject withdrew from the study and second subject got pregnant and was withdrawn, two other subjects still participating in the study did not have ECGs done (which was a protocol violation).) | 25
Completed | 21
Not Completed | 4
Not completed — Pregnancy | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2
Period: Ranolazine
Arm/Group | Placebo
Started (ECG data were available at 1 months in 21 of 25 subjects: one subject withdrew from the study and second subject got pregnant and was withdrawn, two other subjects still participating in the study did not have ECGs done (which was a protocol violation) but they still participated in the period 2. This is why period 2 was started by 23 patients.) | 23
Completed | 18
Not Completed | 5
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: There were 25 subjects that started the study receiving placebo for 1 month.
Arm/Group | All Participants
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 22
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 25
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 25
QTc duration [Mean (Standard Deviation); unit: miliseconds] | 493 (55)

OUTCOME MEASURES:

1. Primary Outcome: Change in QTc Duration at 2 Months
Description: Change in QTc at 2 months on ranolazine vs. at 1 month on placebo. This was prespecified outcome.
Time Frame: 1 month to 2 months
Measure: Mean (Standard Deviation); unit: miliseconds
Groups:
- Placebo: Placebo was administered for 1 month.
- Ranolazine at 2 Months: Ranolazine was administered after 1 month
Arm/Group | Placebo | Ranolazine at 2 Months
Number analyzed (Participants) | 25 | 23
miliseconds | 503 (46) | 497 (47)
Statistical Analysis 1: Comparison: Placebo vs Ranolazine at 2 Months; Test type: Superiority; p = 0.7958, t-test, 2 sided; Paired t-test was used; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-14.1 to 11.0], Standard Deviation 26.8

2. Secondary Outcome: Change in QTc at 6 Months
Description: Change in QTc at 6 months on ranolazine vs. at 1 month on placebo. This was prespecified outcome.
Time Frame: 1 month to 6 months
Measure: Mean (Standard Deviation); unit: miliseconds
Groups:
- Placebo: Placebo administered at first month.
- Ranolazine at 6 Months: Ranolazine was administered for 5 months following 1 month on placebo.
Arm/Group | Placebo | Ranolazine at 6 Months
Number analyzed (Participants) | 23 | 21
miliseconds | 504 (53) | 501 (49)
Statistical Analysis 1: Comparison: Placebo vs Ranolazine at 6 Months; Test type: Superiority; p = 0.3369, t-test, 2 sided; Paired t-test was used; Median Difference (Final Values) = 8.4, 95% CI 2-sided [-9.5 to 26.2], Standard Deviation 35.9

ADVERSE EVENTS:
Time Frame: Adverse events data were collected for 1 month on placebo and for up to 5 months on ranolazine.
Groups:
- Ranolazine: During 5 months on ranolazine following adverse events were reported:
  Ventricular fibrillation successfully treated with shock from implantable cardioverter-defibrillator (n=1) Ventricular fibrillation unsuccessfully treated with shock from implantable cardioverter-defibrillator with subsequent death (n=1) Bundle branch block (n=1) Dizziness/unsteadiness (n=3) Headache (n=1) Constipation (n=1) Hematuria (n=1) Hemorrhoids (n=1)
- Placebo: During 1 month on placebo following adverse events were reported:
  Pregnancy (n=1) Gastritis (n=1) Generalized weakness (n=1)
Arm/Group | Ranolazine | Placebo
All-Cause Mortality (participants affected / at risk) | 1/25 | 0/25
Serious Adverse Events (participants affected / at risk) | 2/25 | 0/25
Other Adverse Events (participants affected / at risk) | 3/25 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=25) | Placebo (N=25)
Ventricular Fibrillation (Cardiac disorders) | 2 (2) | 0 (0) — Ventricular Fibrillation is a life-threatening ventricular arrhythmia.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ranolazine (N=25) | Placebo (N=25)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) — Unsteadiness

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT01648205/Prot_SAP_000.pdf
  • Informed Consent Form (2012-08-15): https://cdn.clinicaltrials.gov/large-docs/05/NCT01648205/ICF_001.pdf